CLINICAL TRIAL: NCT07140081
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled Single-ascending Dose and Multiple-ascending Dose (SAD and MAD) Trial to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of the Isoform-specific AMPK Activator BLX-0871 in Healthy Adults With a Body Mass Index (BMI) of 20 - 35 kg/m2
Brief Title: A Research Study to Evaluate BLX-0871 in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biolexis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BLX-0871-CLN-001
Record Dates: First submitted 2025-08-04; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Normal Healthy Adults
Keywords: BLX-0871; 0871; Obesity; Metabolic disorders; Normal health volunteer
MeSH Terms: conditions — Obesity; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BLX-0871 Oral Dose (Experimental): Participants will receive oral BLX-0871 as a single dose (in Part 1 or 2) or once daily for 7 days (in Part 3).
  Interventions: Drug: BLX-0871
- Placebo to match BLX-0871 (Placebo Comparator): Participants will receive an oral placebo that looks like BLX-0871 but does not contain active drug as a single dose (in Part 1 or 2) or once daily for 7 days (in Part 3).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BLX-0871 — BLX-0871 Single or Multiple doses administered orally as a tablet
  Arms: BLX-0871 Oral Dose
Drug: Placebo — Participants will receive matching placebo of BLX-0871 for each of the oral cohorts.
  Arms: Placebo to match BLX-0871

SUMMARY:
This study will test an oral medicine called BLX-0871, which is being developed to improve metabolic health by activating AMP-activated protein kinase (AMPK), a key regulator of energy balance. The main goal is to see if BLX-0871 is safe and well tolerated when given to healthy adults. The study will also measure how the body processes BLX-0871, including how quickly it is absorbed, how long it stays in the blood, and how it is eliminated. Another objective is to see whether food affects the absorption of BLX-0871. It will also look at how the drug affects the body by looking at markers of AMPK activity.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, first-in-human study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and the effect of food on the PK of BLX-0871, a novel oral small-molecule AMPK activator, in healthy adult volunteers. The study consists of three parts: single ascending dose (SAD), food effect (FE), and multiple ascending dose (MAD) assessments.

Study Rationale and Objectives BLX-0871 is being developed as an oral small-molecule activator of AMP-activated protein kinase (AMPK), a central regulator of energy metabolism. AMPK activation promotes glucose uptake and fatty acid oxidation, supporting potential use in metabolic diseases such as type 2 diabetes and obesity. This first-in-human study is designed to characterize the initial safety profile, define the PK properties of BLX-0871, evaluate preliminary PD biomarkers of metabolic activity, and determine the impact of a high-fat meal on oral absorption.

Study Design Overview The study will enroll approximately 76 healthy adults across three sequential parts.

Part 1: Single Ascending Dose (SAD) This is a randomized, double-blind, placebo-controlled, sequential SAD study in up to four cohorts (approximately 8 participants per cohort; 6 active, 2 placebo). Doses will escalate sequentially following review of blinded safety, tolerability, PK, and PD data by a Safety Review Committee (SRC). A sentinel dosing approach will be used for each cohort (1 active, 1 placebo) prior to dosing the remainder of the cohort. Participants will be confined in the clinical research unit (CRU) for approximately 4 days for safety monitoring and PK/PD blood sampling, with an end-of-study (EOS) visit on Day 8. SAD data will inform dose selection for the FE and MAD parts of the study.

Part 2: Food Effect (FE) This is an open-label, randomized, 2-period, 2-sequence crossover study designed to evaluate the effect of a high-fat, high-calorie meal on the PK of a single oral dose of BLX-0871. A single cohort of 12 participants will receive BLX-0871 under both fasted and fed conditions, with a 7-day washout between doses. Participants will be confined for approximately 4 days in each period, with safety, PK, and PD assessments performed throughout. The SRC may adjust the washout interval or timing of assessments based on PK results from the SAD cohorts to ensure adequate elimination between periods.

Part 3: Multiple Ascending Dose (MAD) This is a randomized, double-blind, placebo-controlled, sequential MAD study in up to four cohorts (approximately 8 participants per cohort; 6 active, 2 placebo). Participants will receive BLX-0871 or placebo orally once daily for 7 days. Participants will be confined from Day -1 through approximately Day 10 for dosing, safety assessments, and PK/PD sampling, with an EOS visit on Day 14. Dose escalation to subsequent MAD cohorts will occur following review of blinded safety, PK, and PD data by the SRC.

Safety Monitoring Safety will be evaluated throughout the study by monitoring adverse events (AEs), clinical laboratory tests, vital signs, 12-lead electrocardiograms (ECGs), echocardiograms, and physical examinations. Sentinel dosing and SRC reviews between cohorts are incorporated to minimize risk.

Pharmacokinetic and Pharmacodynamic Assessments Blood samples will be collected to characterize single- and multiple-dose PK parameters of BLX-0871, including maximum concentration (Cmax), time to maximum concentration (Tmax), area under the curve (AUC), half-life (t½), and apparent clearance. PD assessments will evaluate exploratory biomarkers of metabolic activity, including fasting glucose, insulin, free fatty acids, and ketones. These data will provide early evidence of biological activity and support dose selection for future studies.

Dose Escalation and Cohort Progression The SRC will review cumulative safety, tolerability, PK, and PD data after each cohort before escalating to the next dose level. The number of cohorts may be reduced based on emerging data. The FE and MAD parts may proceed in parallel with later SAD cohorts once predefined safety criteria are met.

The results of this study will provide the initial clinical safety, PK, and PD profile of BLX-0871, including a preliminary assessment of food effect, to support future clinical development in populations with metabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, 18-65 years, BMI 20-35 kilograms/meter² (kg/m²), weight ≥50 kilograms (kg).
* Normal or clinically acceptable labs, vital signs
* HbA1c <6.5%, non-fasting glucose 4.0-7.8 milimol/Liter (mmol/L)
* Willing to follow contraception requirements, avoid alcohol, nicotine, and blood donation per protocol, and comply with all study visits and procedures.

Exclusion Criteria:

* History of diabetes, clinically significant cardiovascular, hepatic, renal, gastrointestinal, psychiatric, or neurologic disease, or abnormal labs/Echocardiograms (ECG) deemed clinically relevant.
* Prior gastrointestinal (GI) surgery affecting absorption (e.g., gastric bypass) or chronic GI disorders.
* History or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia type 2 (MEN2); malignancy within 5 years (except treated basal cell or in situ cervical cancer).
* History of severe allergic reactions, seizures, or psychiatric hospitalization; positive drug, alcohol, or cotinine test.
* Use of prescription drugs, Over the counter (OTC) /herbal supplements
* Participation in another clinical trial or blood donation within 30 days (or 5 half-lives of prior drug).
* Any condition or history that may compromise safety, study conduct, or compliance, in the opinion of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experienced Adverse Events (AEs) | From first dose through End of Study (up to ~28 days per participant)
  The safety and tolerability of oral BLX-0871 administration will be evaluated based on the incidence of adverse effects in subjects, as assessed according to CTCAE v5.0. The number of participants who experience an AE will be reported.
Number of participants who experienced Serious Adverse Events (SAEs) | From first dose through End of Study (up to ~28 days per participant)
  The safety and tolerability of oral BLX-0871 administration will be evaluated based on the incidence of SAE in subjects, as assessed according to CTCAE v5.0. The number of participants who experience a SAE will be reported.
Number of participants who experienced Treatment-Related Adverse Avents (TRAEs) | From first dose through End of Study (up to ~28 days per participant)
  The safety and tolerability of oral BLX-0871 administration will be evaluated based on the incidence of TRAEs in subjects, as assessed according to CTCAE v5.0. The number of participants who experience a TRAE will be reported.

SECONDARY OUTCOMES:
Assess maximum observed drug concentration (Cmax) | Up to 14 days after last dose in each cohort
  Evaluate the relative bioavailability of BLX-0871 in single, food effect, and multiple ascending doses in healthy adults
Assess time to maximum concentration (Tmax) | Up to 14 days after last dose in each cohort
  Evaluate the relative bioavailability of BLX-0871 in single, food effect, and multiple ascending doses in healthy adults
Assess the area under the concentration-time curve from time 0 to infinity (AUCinf) | Up to 14 days after last dose in each cohort
  Evaluate the relative bioavailability of BLX-0871 in single, food effect, and multiple ascending doses in healthy adults
Assess the area under the concentration curve from time 0 to the last quantifiable concentration (AUClast) | Up to 14 days after last dose in each cohort
  Evaluate the relative bioavailability of BLX-0871 in single, food effect, and multiple ascending doses in healthy adults
Assess half-life (t½) plasma concentration | Up to 14 days after last dose in each cohort
  Evaluate the relative bioavailability of BLX-0871 in single, food effect, and multiple ascending doses in healthy adults
Serum fructosamine | Up to 14 days after last dose in each cohort
  Evaluate the effect of single and multiple oral doses of BLX-0871 on serum fructosamine levels
Plasma levels of phosphorylated AMPK (pAMPK) and total AMPK | Up to 14 days after last dose in each cohort
  Evaluate the effect of multiple oral doses of BLX-0871 on plasma levels of phosphorylated AMPK (pAMPK) and total AMPK
Plasma levels of phosphorylated acetyl-CoA carboxylase ACC (pACC) and total ACC | Up to 14 days after last dose in each cohort
  Evaluate the effect of multiple oral doses of BLX-0871 on plasma levels of levels of phosphorylated acetyl-CoA carboxylase ACC (pACC) and total ACC

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network St Kilda Road, Melbourne, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No